CLINICAL TRIAL: NCT00909259
Title: Feasibility Study to Determine the Effects of Phrenic Nerve Stimulation in Patients With Periodic Breathing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Respicardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-Feasibility
Record Dates: First submitted 2009-05-21; First posted 2009-05-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Sleep Disordered Breathing; Cheyne-Stokes Respiration; Sleep Apnea
Keywords: Sleep Disordered Breathing; Periodic Breathing; Cheyne-Stokes Respiration; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Cheyne-Stokes Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phrenic Stimulation (Experimental)
  Interventions: Device: Phrenic stimulation device

INTERVENTIONS:
Device: Phrenic stimulation device — In Stage 1, a stimulation lead will be introduced via standard access methods and positioned to provide stimulation. A second lead may also be placed for sensing purposes. The proximal portions of the implanted lead(s) will remain externalized such that stimulation and observation can be made using external stimulation and recording equipment. Study subjects will be observed and stimulation will be performed for up to 2 nights of sleep in a clinically supported environment. In Stage 2, a stimulation device and lead will be permanently implanted.

SUMMARY:
The purpose of this feasibility study is to determine the effect of stimulating the phrenic nerve to treat periodic breathing (a pattern of breathing characterized by hyperpneas followed by hypopneas or apneas). Clinically, these physiologic events translate into sleep fragmentation, excessive daytime sleepiness, reduced exercise capacity, and possibly ventricular arrhythmias.

Stage 1 of the study is acute in nature, such that subjects will undergo the placement of a stimulation lead, followed by assessment of stimulation of the phrenic nerve using the lead for up to 2 nights of sleep. A sensing lead may also be placed during the initial implant procedure. Observational data will be obtained and stimulation provided using an externalized system connected to the study leads. Following the study, all investigational components will be removed from the patient.

Stage 2 of the study is being conducted at one of the participating sites to determine the initial safety of chronic stimulation of the phrenic nerve in a limited number of patients with sleep disordered breathing. It is anticipated that data obtained in this feasibility study will show that the proposed intervention can modify respiration with a low incidence of adverse effects. The results of this trial are intended to be used to develop a subsequent protocol for a multi-center study of chronic phrenic nerve pacing.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient has a demonstrated history of periodic breathing (symptoms may include sleep fragmentation, as reported by patient or as witnessed by another person, night arousal after apneic episodes, reduced exercise capacity, and daytime sleepiness)
* Patient is expected to be able to tolerate the procedure and remain clinically stable for the duration of the study (e.g. the subject is able to lie down long enough to insert the lead(s) without shortness of breath and the subject is able to tolerate instrumentation during study).
* Patient or their legal representative is willing and able to sign an IRB/MEC approved informed consent (and a privacy protection authorization in the United States)

Exclusion Criteria:

* Baseline oxygen saturation less than or equal to 90% on a stable FIO2
* Evidence of phrenic nerve palsy
* Temperature > 38.0 degrees Celsius
* Inability to place catheter (e.g. previously known coagulopathy, distorted anatomy, etc.)
* Patient is currently enrolled in another study that may confound the results of this study
* Patient for whom informed consent cannot be obtained
* Patient who is pregnant or of child bearing potential without a negative pregnancy test within 10 days of the study procedure
* Patients implanted with a pacemaker, implantable defibrillator, or cardiac resynchronization device who are unable to tolerate turning off the device for the duration of the system testing procedure (based on medical judgment)
* Patients with severe COPD (per GOLD scale)
* Patients with a history of myocardial infarction within 6 months prior to the study
* Patients with unstable angina
* Patients who are intolerant of or allergic to contrast dye
* Patients who are contraindicated for <1mg of steroid (on the stimulation lead).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary goal of this feasibility study is to show an acute improvement in respiration. | Acute (up to 2 nights of sleep)
The primary safety endpoint of the study is the absence of adverse events related to stimulation that result in hospitalization, the prolongation of an existing hospitalization, or death of the patient. | Acute (up to 2 nights of sleep) plus post-operative assessment at one week (5-10 days) or until resolution of an observed adverse event.

SECONDARY OUTCOMES:
Characterization of chronic safety of stimulating the phrenic nerve (Stage 2 of study). | 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Ohio Heart Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
- Jiangsu Province Hospital, Nanjing, China
- Polish Military Hospital, Wroclaw, Poland

REFERENCES:
- [Derived] Zhang XL, Ding N, Wang H, Augostini R, Yang B, Xu D, Ju W, Hou X, Li X, Ni B, Cao K, George I, Wang J, Zhang SJ. Transvenous phrenic nerve stimulation in patients with Cheyne-Stokes respiration and congestive heart failure: a safety and proof-of-concept study. Chest. 2012 Oct;142(4):927-934. doi: 10.1378/chest.11-1899. PMID 22302299
- [Derived] Ponikowski P, Javaheri S, Michalkiewicz D, Bart BA, Czarnecka D, Jastrzebski M, Kusiak A, Augostini R, Jagielski D, Witkowski T, Khayat RN, Oldenburg O, Gutleben KJ, Bitter T, Karim R, Iber C, Hasan A, Hibler K, Germany R, Abraham WT. Transvenous phrenic nerve stimulation for the treatment of central sleep apnoea in heart failure. Eur Heart J. 2012 Apr;33(7):889-94. doi: 10.1093/eurheartj/ehr298. Epub 2011 Aug 19. PMID 21856678